CLINICAL TRIAL: NCT02019043
Title: Enhanced Syphilis Screening Among HIV-positive Men (ESSAHM): Evaluation of a Clinic-based Intervention
Brief Title: Evaluation of Enhanced Syphilis Screening Among HIV-positive Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); Toronto General Hospital (Other); Ontario HIV Treatment Network (Network); The Ottawa Hospital (Other); Sunnybrook Health Sciences Centre (Other); Ontario Agency for Health Protection and Promotion (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MOP 130440
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Syphilis Serodiagnosis

STUDY DESIGN:
Intervention Model Description: Note: Although the trial period and recruitment is complete, data entry is ongoing. Completion of data entry is anticipated for August 2018.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Syphilis testing with routine HIV bloodwork (Experimental): The intervention condition will be implemented as standing orders for syphilis serology whenever patients undergo their standard battery of follow-up bloodwork, i.e., when there is an order for HIV viral load or CD4 cell count.
  Interventions: Other: Syphilis testing with routine HIV bloodwork
- Current care practice (No Intervention): The control condition will remain the current care practice, which is generally opportunistic screening or diagnostic testing for those presenting with signs/symptoms or who report sexual risk behaviour.

INTERVENTIONS:
Other: Syphilis testing with routine HIV bloodwork — The intervention condition will be implemented as standing orders for syphilis serology whenever patients undergo their standard battery of follow-up bloodwork, i.e., when there is an order for HIV viral load or CD4 cell count. It is standard practice for HIV patients to undergo such tests every 3-6 months. We anticipate that the change in practice will be straightforward, involving minimal training of clinic staff. Team members who are physicians at these clinics will guide the specific approach that will be appropriate and sustainable for their setting. Options are quite simple. They include pre-printing a checkmark for 'syphilis serology' onto existing pre-printed requisitions for routine bloodwork; addition of the serology request form to the routine blood work package; or programming 'syphilis serology' into existing computerized routine order sets.
  Arms: Syphilis testing with routine HIV bloodwork

SUMMARY:
This study aims to enhance syphilis testing among HIV-positive men who have sex with men (MSM), so that more men will undergo testing, they will test more often, and more cases will be treated early. The intervention will combine syphilis tests with the standard HIV blood tests that are routinely done every 3-6 months for persons in care at hospital-based HIV clinics in Toronto and Ottawa, Canada.

DETAILED DESCRIPTION:
A clinic-based intervention to incorporate syphilis testing with routine HIV bloodwork among HIV-positive men who have sex with men (MSM) attending 4 hospital-based HIV clinics in Toronto and Ottawa will be conducted. The objectives are to determine to what degree the intervention: (1) increases the detection rate of untreated syphilis; (2) increases the proportion of men who undergo syphilis testing at least annually (increased screening coverage); (3) reduces the interval between syphilis tests (increased screening frequency); and (4) reaches men at highest risk according to sexual behaviours. The main hypotheses are that the intervention will increase screening coverage to a minimum of 85% of men undergoing syphilis testing annually, increase screening frequency to a median of 3 tests per person per year, and increase the case detection rate by 75% or more.

The design of this study is a cluster-randomized controlled trial with stepped wedge design that will gradually introduce the intervention across clinics. This pragmatic approach incorporates a concurrent comparison group, allows for assessment of time trends, will be well-powered, and will generate more generalizable results due to its inclusion of multiple clinics. The intervention will be operationalized as standing orders for syphilis serology when there is an order for HIV viral load and/or CD4 cell count. Data sources include (1) syphilis tests submitted to the Public Health Ontario Laboratory; (2) a standardized clinical worksheet and medical chart review to validate diagnoses for screen test positives; and (3) data collected from a subset of patients via their participation in the ongoing Ontario HIV Treatment Network (OHTN) Cohort Study. The latter follows adults in HIV care and collects data using chart reviews and annual face-to-face interviews including measures of sexual behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Male HIV patients
* Must be attending at least one of the four participating hospital-based HIV outpatient clinics

Exclusion Criteria:

* Women

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3895 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in rate of detection of new, previously untreated syphilis cases | At 30 months
  We will use a cluster-randomized controlled trial (CRCT) using a stepped wedge design that will gradually introduce the intervention across four clinics. Each clinic will be randomized to one of the four roll-out periods, and will have at minimum one 6-month control period and one 6-month intervention period. The main hypothesis to be tested is H0: θ=0 versus Ha: θ= θa where θ represents the increase in the case detection rate due to the intervention and θa represents a 75% increase over the baseline rate.

SECONDARY OUTCOMES:
Change in screening coverage | At 30 months
  Proportion tested for syphilis at least once per year
Change in screening frequency | At 30 months
  Number of times tested for syphilis, per year.

OTHER OUTCOMES:
Direct and indirect costing of each additional screen-detected syphilis diagnosis | Month 30
  Costs will include inpatient services (initial screening and follow-up management costs), drug costs, syphilis test kits and technician time.

CONTACTS AND LOCATIONS:
Overall Officials: Ann N Burchell, PhD, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] MacKinnon KR, Grewal R, Tan DH, Rousseau R, Maxwell J, Walmsley S, MacPherson PA, Rachlis A, Andany N, Mishra S, Allen VG, Burchell AN. Patient perspectives on the implementation of routinised syphilis screening with HIV viral load testing: Qualitative process evaluation of the Enhanced Syphilis Screening Among HIV-positive Men trial. BMC Health Serv Res. 2021 Jun 30;21(1):625. doi: 10.1186/s12913-021-06602-1. PMID 34193138
- [Derived] Burchell AN, Tan DHS, Grewal R, MacPherson PA, Walmsley S, Rachlis A, Andany N, Mishra S, Gardner SL, Raboud J, Fisman D, Cooper C, Gough K, Maxwell J, Rourke SB, Rousseau R, Mazzulli T, Salit IE, Allen VG. Routinized Syphilis Screening Among Men Living With Human Immunodeficiency Virus: A Stepped Wedge Cluster Randomized Controlled Trial. Clin Infect Dis. 2022 Mar 9;74(5):846-853. doi: 10.1093/cid/ciab582. PMID 34175944
- [Derived] Burchell AN, Allen VG, Grewal R, MacPherson PA, Rachlis A, Walmsley S, Mishra S, Gardner SL, Raboud J, Cooper C, Gough K, Rourke SB, Rousseau R, Salit I, Tan DH. Enhanced syphilis screening among HIV-positive men (ESSAHM): a study protocol for a clinic-randomized trial with stepped wedge design. Implement Sci. 2016 Jan 16;11:8. doi: 10.1186/s13012-016-0371-0. PMID 26772390